CLINICAL TRIAL: NCT06623565
Title: Multimodal Image-guided Resection of IDH Wildtype Glioblastoma and Grade IV IDH-mutant Astrocytoma
Brief Title: Extensive Resection of Malignant Brain Tumors Using Advanced Imaging Techniques
Acronym: NEXTFRONTIER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, dr. Niels Verburg, Neurosurgeon, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.0020; CCA2021-5-27 (Other Grant/Funding Number: Cancer Center Amsterdam)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma; Astrocytoma, IDH-Mutant, Grade 4
Keywords: multimodal imaging; high grade glioma; glioblastoma; supramarginal; resection; surgery
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Supramarginal resection using combination of ADC MRI and FET PET
  Interventions: Procedure: Multimodal image-guided resection

INTERVENTIONS:
Procedure: Multimodal image-guided resection — Supramarginal resection using combination of ADC MRI and FET PET

SUMMARY:
Rationale: Patients with IDH-wildtype glioblastoma or grade IV IDH-mutant astrocytoma have a very poor prognosis despite standard treatment consisting of surgery, radiotherapy, and chemotherapy. Diffuse infiltration of the brain by the tumor is thought to be one of the main causes of this therapy-resistance. In order to improve the surgical treatment, tumor regions with lower infiltration percentages need to be identified and resected during surgery, a so-called supramarginal resection. Currently, pre-operative T1 contrast enhanced weighted (T1c) MRI is used to identify the tumor for resection. We recently found the combination of apparent diffusion coefficient MRI and O-(2-[ 18F]fluoroethyl-)-L-tyrosine positron emission tomography (ADC/FET) to be significantly more accurate than T1c MRI alone in the detection of tumor infiltration. This makes ADC/FET a suitable candidate to guide supramarginal resection. Since FET PET is not as accessible and widely available as MRI, identification of an MRI based alternative could result in a more widespread implementation. Amide proton transfer chemical exchange saturation transfer (APT-CEST) MRI is a novel potential alternative for FET PET, since both measures are related to protein content.

Objective: In this project we aim to develop a safe and effective technique for ADC/FET guided resection of IDH-wildtype glioblastoma and grade IV IDH-mutant astrocytoma. The safety concerns neurological deficits and time to start of adjuvant therapy, while the effectiveness is aimed at the extent of resection. Our secondary aim is to evaluate the diagnostic accuracy of APT-CEST MRI and to assess whether APT-CEST MRI can serve as an alternative for FET PET for the detection of tumor infiltration.

Study design: prospective observational intervention study

Study population: 30 patients with clinical and radiological diagnosis of an untreated high grade glioma (suspected for glioblastoma (IDH wildtype) or grade IV astrocytoma (IDH mutant)), who are eligible for a supramarginal surgical resection and adjuvant treatment according two neurosurgeons in consensus and who are in relatively good condition (Karnofsky Performance Score (KPS) ≥70).

Intervention (if applicable): supramarginal ADC/FET-guided resection. To make sure that the standard treatment is always guaranteed, T1c MRI abnormalities will be included in the surgical target.

Main study parameters/endpoints: the main study endpoint is the optimization of ADC/FET-guided resection. Volumetric and percentual extent of resection, as measured with MRI and PET imaging, combined with surgery-induced morbidity will be used as outcome parameters. The secondary study parameters will be the histopathology-based diagnostic accuracy of APT-CEST MRI in comparison with FET PET, cognitive performance over time and progression free survival.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: participants will undergo pre- and postoperative MRI scanning. This is also part of regular clinical care, except there are additional MRI sequences including APT CEST in the pre-operative and pre-radiotherapy MRI. There are no risks associated with MRI acquisition after MRI safety screening. Participants will furthermore undergo a pre- and postoperative FET PET. The risks associated with PET scanning are limited, and the radiation burden will remain below 10 mSv (ICRP62 category intermediate risk (level IIb)). During surgery, biopsies are performed from areas that will be resected, so these biopsies will not introduce any extra risk. A potential benefit is the possibility of the removal of more tumor tissue. A potential risk is the additional removal of healthy brain tissue with the risk of neurological damage, which is controlled by pre- and intraoperative techniques such as visualization of white matter tracts and mapping (both asleep and awake) of critical functions such as language and control of strength.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* New clinical and radiological suspected diagnosis of IDH-wildtype glioblastoma or grade IV IDH-mutant astrocytoma
* Visible FET PET uptake in the tumor as assessed by the nuclear physician
* Indication for a surgical resection and adjuvant treatment according to the neuro oncology multidisciplinary meeting
* Eligible for a supramarginal resection according to two neurosurgeons in consensus
* Karnofsky Performance Score (KPS) ≥ 70.

Exclusion Criteria:

* Previous brain surgery or cranial radiotherapy
* No significant other brain pathology, in the opinion of the PI or designee, such as multiple sclerosis, neurodegenerative disease, stroke
* Tumor located infratentorially or in the spinal cord
* Lack of adequate social or family support needed for adherence to the further postoperative therapeutic regimen
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Extent of resection | within 4 weeks after surgery
  Volumetric and percentual on pre-radiotherapy PET-MRI
Neurological functioning | 3 months after surgery
  Neurological Assessment in Neuro-Oncology (NANO) score

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided